CLINICAL TRIAL: NCT02893111
Title: Single-center, Open Label Trial of Bortezomib as add-on Treatment in Relapsing Neuromyelitis Optica Spectrum Disorder
Brief Title: Efficacy and Safety of Bortezomib as add-on Treatment in Relapsing Neuromyelitis Optica Spectrum Disorder
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: Tianjin Medical University General Hospital (Other)
Responsible Party: Principal Investigator, Fu-Dong Shi, Director of Neurology, Tianjin Medical University General Hospital
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: IRB2016-YX-021
Record Dates: First submitted 2016-08-27; First posted 2016-09-08 (Estimated); Last update posted 2024-04-11 (Actual); Status verified 2024-04

CONDITIONS: Neuromyelitis Optica Spectrum Disorder
Keywords: neuromyelitis optica spectrum disorders; Bortezomib; Velcade; Proteasome inhibitor
MeSH Terms: conditions — Neuromyelitis Optica | interventions — Bortezomib

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (1):
- Bortezomib (Velcade) (Experimental): A proteasome inhibitor
  Interventions: Drug: Bortezomib

INTERVENTIONS:
Drug: Bortezomib — Bortezomib will be subcutaneously applicated in 4 treatment cycles with 4 injections of 1 mg Bortezomib /m2 body surface per cycle
  Other Names: Velcade

SUMMARY:
Neuromyelitis Optica Spectrum Disorders (NMOSD) is characterized by the pathogenic anti-AQP4 antibody, which can be produced by specific plasma cells. The patients who are not responsive to rituximab treatment may be due to the presence of short-lived and long-lived plasma cells. Previous studies confirmed that the proteasome inhibitor bortezomib (Velcade®, approved for therapy of multiple myeloma) eliminated both plasmablasts and plasma cells by activation of the terminal unfolded protein response. Treatment with bortezomib may help deplete plasma cells producing auto-antibodies. Therefore, the rationale for using bortezomib in NMOSD is in that bortezomib may help eliminate autoreactive plasma cells and reduce anti-AQP4 antibodies titers. It is noted that bortezomib may protect astrocytes from NFκB-dependent inflammatory damage in early events in NMOSD pathogenesis.

The purpose of this study is to determine if the drug bortezomib contributes to reduce the average relapsing rates (ARRs) and alleviate neurological disability in NMOSD patients.

DETAILED DESCRIPTION:
It has been shown in some scientific studies that the the antibody marker specific for neuromyelitis optica spectrum disorders (NMOSD), known as AQP4-IgG, causes inflammation in brain tissues by activating NF-κB pathway. Bortezomib has already been shown to be effective in systemic lupus erythematosus (SLE).

The overall objective is to assess the efficacy and safety of bortezomib as add-on therapy to oral steroids,azathioprine or others for treatment of relapsing NMOSD, which have not reduced average relapsing rate (ARR) effectively.

The primary (most important) objectives of this study are to determine:

Whether bortezomib reduces relapse frequency in patients with relapsing NMO. The number of attacks during the one year treatment period will be compared to the number of attacks that occurred prior to initiation of bortezomib treatment.

The secondary objectives are to determine:

The safety profile of bortezomib in patients with NMO. Whether bortezomib maintains or improves walking, visual function and quality of life as measured by a variety of established disability scales. We will also assess the severity of an individual attack and the degree of recovery.

Depending on our preliminary investigations we may evaluate patient cerebrospinal fluid in the laboratory to see how effective eculizumab is at getting into the cerebrospinal fluid from the blood stream, and to see if the drug reverses the biological effects of the NMO-IgG antibody.

ELIGIBILITY:
Inclusion Criteria:

* Age ≥18 years
* Diagnosis of NMOSD, as defined by 2015 criteria OR NMOSD seropositive spectrum disorder (Recurrent ON or longitudinally extensive transverse myelitis (LETM)). All patients must be NMO-IgG seropositive.
* Clinical evidence of at least 2 relapses in last 6 months or 3 relapses in the last 12 months (with at least 1 relapse occurring in the preceding 6 months)
* The B cell count must be normal (5-20% of total lymphocytes) in subjects before administration of bortezomib
* Provision of written informed consent to participate in the study
* Corrected visual acuity 20/100 or better in at least one eye; otherwise, last attack was myelitis and only attacks of myelitis are outcomes
* Ambulatory (with or without walker); otherwise, last attack was optic neuritis and only attacks of optic neuritis are outcomes

Exclusion Criteria:

* Current evidence or known history of clinically significant infection (HSV, VZV, CMV, EBV, HIV, Hepatitis viruses, Syphilis, etc)
* Pregnant, breastfeeding, or child-bearing potential during the course of the study
* Patients will not participate in any other clinical therapeutic study or will not have participated in any other experimental treatment study within 30 days of screening
* Patients with a history of splenectomy, because of a potential increased risk of developing meningococcal infection
* Participation in another interventional trial within the last 3 months
* Pre-existent sensory or motor polyneuropathy ≥ degree 2 (NCI CTC AE criteria), within 14 days before screening
* Heart or kidney insufficiency
* Tumor disease currently or within last 5 years
* Clinically relevant liver, kidney or bone marrow function disorder

Ages: 18 Years to 75 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 5 (Actual)
Dates: Start 2015-12; Primary Completion 2016-12-25 (Actual); Study Completion 2017-01-31 (Actual)

PRIMARY OUTCOMES:
Annual relapse rate (ARR) of NMOSD Attacks | Baseline, after 12 months of initial treatment
  Compare annual relapse rate before and one year after initial Bortezomib administration

SECONDARY OUTCOMES:
Number of Participants with Adverse Events | Baseline, 12 months
  All adverse events and side effects related to this drug will be recorded
Change in Expanded Disability Status Scale (EDDS) Score | Baseline, 12 months
  The EDSS is an ordinal clinical rating scale ranging from 0 (normal neurologic examination) to 10 (death) in half-point increments.
Timed 25-foot Walk | Baseline, 12 months
  The Timed 25-Foot Walk test is a quantitative measure of lower extremity function
Number of Subjects With Change in Visual Acuity in at Least One Eye by at Least One Point | Baseline, 12 months
  Visual acuity was measured using the the visual acuity subscale of the opticospinal impairment score (OSIS) for Exacerbations. This subscale ranges from 0 (normal) to 8 (no light perception).
MRI brain and spine | Baseline, 12 months
  MRIs will be analyzed for counting the numbers of new lesions by T2 hyper-intensity in the brain, spinal cord and optic nerve (minimal number is 0), and the volume of T1 post-contrast enhancement (minimal volume is 0 cm3).
Retinal nerve fiber layer (RNFL) | Baseline, 12 months
  Compared RNFL before and one year after initial Bortezomib administration
Cognition | Baseline, 12 months
  Compare cognition questionnaire scale before and one year after initial Bortezomib administration
Immunological assessments | Baseline, 12 months
  Compare Ig subclasses (serum IgG1,IgG2, IgG3 and IgG4 concentrations by mg/dL), anti-aquaporin4-ab (measured by FIPA nmol/L and FACS assay titre), cytokine kinetics (measured by ELISA assay titre), relevant plasma cells depletion (number of circulating cells measured by count/μL ) before and one year after initial Bortezomib administration

CONTACTS AND LOCATIONS:
Locations (1):
- Tianjin Medical University General Hospital, Tianjin, Tianjin Municipality, China

IPD SHARING:
Plan to Share IPD: No